CLINICAL TRIAL: NCT03013348
Title: Automated Identification of Psychogenic Nonepileptic Seizures
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brain Sentinel (Other)
Responsible Party: Sponsor
Other Study IDs: NES-1.5-09.2016
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Convulsion, Non-Epileptic
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Adults (22-99),: Male or female subject between the ages of 22-99, previously admitted to the Medical University of South Carolina for inpatient vEEG monitoring in the MUSC Epilepsy Monitoring Unit with at least one PNES was recorded during that admission. Validation of Brain Sentinel's sEMG Post-processing algorithm will involve prospective evaluation of at least 30 PNES events in this group.
  Interventions: Device: Brain Sentinel's sEMG Post-processing algorithm
- Adolescents (13-21): Male or female subject between the ages of 13-21, previously admitted to the Medical University of South Carolina for inpatient vEEG monitoring in the MUSC Epilepsy Monitoring Unit with at least one PNES was recorded during that admission. Validation of Brain Sentinel's sEMG Post-processing algorithm will involve prospective evaluation of at least 30 PNES events in this group.
  Interventions: Device: Brain Sentinel's sEMG Post-processing algorithm
- Children (2-12): Male or female subject between the ages of 2-12, previously admitted to the Medical University of South Carolina for inpatient vEEG monitoring in the MUSC Epilepsy Monitoring Unit with at least one PNES was recorded during that admission. Validation of Brain Sentinel's sEMG Post-processing algorithm will involve prospective evaluation of at least 30 PNES events in this group.
  Interventions: Device: Brain Sentinel's sEMG Post-processing algorithm

INTERVENTIONS:
Device: Brain Sentinel's sEMG Post-processing algorithm — Brain Sentinel has developed a post processing method that identifies sEMG signals (recorded from the biceps brachii or as muscle artifact in electroencephalography [EEG] recordings) that are pathognomonic for PNES activity.

SUMMARY:
A retrospective validation study of a post-processing method intended to identify psychogenic nonepileptic seizures

DETAILED DESCRIPTION:
This is a validation study of a post-processing method intended to identify psychogenic nonepileptic seizures by analysis of surface electromyographic (sEMG) artifact previously recorded during routine video-electroencephalographic (vEEG) monitoring

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study if the following criteria apply.

* Subject was previously admitted to the Medical University of South Carolina for inpatient vEEG monitoring in the MUSC Epilepsy Monitoring Unit and at least one PNES was recorded during that admission.
* Male or female between the ages of 2-99
* Can understand and sign written informed consent, or will have a parent or a legally authorized representative (LAR) who can do so, prior to the performance of any study assessments

Exclusion Criteria:

* No exclusion criteria have been established for this study.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects previously admitted to the Medical University of South Carolina for inpatient vEEG monitoring in the MUSC Epilepsy Monitoring Unit with at least one PNES recorded during that admission.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
> 70% sensitivity of a post processing method for classification of psychogenic nonepileptic seizures in sEMG artifact captured during vEEG recordings as compared to vEEG interpretation by a panel of three independent Neurologists. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Halford, MD, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: No